CLINICAL TRIAL: NCT07158619
Title: Evaluation of the Acquisition of Sustained Unresponsiveness to Cashew Nut Protein Following Oral Allergen-Specific Immunotherapy - Long-Term Follow-Up of Patients From the RCT "Efficacy of Cashew Nut Protein Immunotherapy: A Protocol of a Single-Center Randomized Controlled Trial in the Pediatric Population" (NCT06328504)
Brief Title: Sustained Unresponsiveness (SU) to Cashew Nut Protein Following Oral Allergen-Specific Immunotherapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KB/61/2025
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Food Allergy in Children
Keywords: food allergy, oral immunoteraphy, cashew nut allergy,
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintenance dose of cashew nut protein (1200mg) for 8 months (Experimental): Patients assigned to the experimental group in the first part of the study (RCT) will continue OIT with the maintenance dose of cashew nut protein (1200mg) for the next 8 months.
  Interventions: Dietary Supplement: OIT with cashew nut protein
- Immunotherapy initiated after one year of cashew nut avoidance (Experimental): Patients assigned to the control group in the first part of the study, after one year on a cashew nut elimination diet, will begin immunotherapy following the protocol used in the first part of the study (RCT). Upon completion of this initial phase, they will continue immunotherapy for an additional 8 months.
  Interventions: Dietary Supplement: OIT with cashew nut protein

INTERVENTIONS:
Dietary Supplement: OIT with cashew nut protein — After 8 months of continued oral immunotherapy (OIT) with cashew nuts, patients will undergo hospital-based assessments, including skin prick testing, laboratory evaluations, and an open Oral Food Challenge (OFC) to assess desensitization. Patients who had a negative OFC after 3 months in the initial phase-confirming desensitization-will skip the pre-break OFC and proceed directly to the next stage. Following a 4-week interruption in OIT, patients will return for a final hospital visit, during which a concluding OFC will be conducted to evaluate sustained unresponsiveness. Additional laboratory tests and skin prick testing will also be performed during this visit.

SUMMARY:
This study is a long-term follow-up of participants from the randomized controlled trial (RCT) "Efficacy of Cashew Nut Protein Immunotherapy: A Protocol of a Single-Center Randomized Controlled Trial in the Pediatric Population", NCT06328504. At the end of the original RCT all participants will undergo an open Oral Food Challenge (OFC) to assess desensitization after 3 months on the maintenance dose of OIT. Patients who have completed the first part of the study will be invited to the current part of the project:

* First arm (initial experimental group) - patients will continue oral immunotherapy (OIT) with cashew nut protein (1200mg) for the next 8 months (+/- 3 weeks).
* Second arm (initial control group - one year on a cashew nut elimination diet) - patients will begin OIT following the protocol used in the first part of the study (RCT). Upon completion of this initial phase, they will continue immunotherapy for an additional 8 months (+/- 3 weeks).

After an additional 8 months (+/- 3 weeks) of OIT, all study participants will undergo a 4-week cessation of treatment, followed by an open Oral Food Challenge (OFC) to assess the development of sustained unresponsiveness (SU).

DETAILED DESCRIPTION:
Oral immunotherapy (OIT) is currently recognized as the most effective disease-modifying intervention for IgE-mediated food allergies. The therapeutic objectives of OIT encompass two distinct immunologic outcomes: desensitization and sustained unresponsiveness (SU).

Desensitization refers to a reversible state of increased clinical tolerance to the allergen, dependent on continuous antigen exposure. In contrast, sustained unresponsiveness-considered the optimal endpoint-describes the maintenance of non-reactivity to the allergen following a defined period of OIT discontinuation.

The present study constitutes a long-term follow-up of participants previously enrolled in the randomized controlled trial (RCT) "Efficacy of Cashew Nut Protein Immunotherapy: A Protocol of a Single-Center Randomized Controlled Trial in the Pediatric Population", NCT06328504. Participants who completed the initial treatment phase will be invited to participate in this extended evaluation.

Study Procedures

Following an additional 8 months (±3 weeks) of continued cashew nut protein OIT, eligible participants will undergo a comprehensive in-hospital evaluation, including:

Skin prick testing (SPT) with commercial extracts of peanut, walnut, hazelnut, pistachio, cashew, almond, and native tests with cashew flour, peanut butter, and fresh nuts listed above

Laboratory assessments (e.g., specific IgE, IgG4), and

A standardized open oral food challenge (OFC) to cashew nut protein to assess clinical desensitization.

Participants who demonstrated confirmed desensitization (i.e., negative OFC) after 3 months of OIT during the initial trial phase will proceed to the next phase of the study protocol without repeating an OFC prior to OIT cessation. Only those with previously confirmed desensitization will be eligible for assessment of sustained unresponsiveness.

Following a 4-week discontinuation period (i.e., OIT treatment break), these participants will undergo a second OFC to evaluate sustained unresponsiveness to cashew nut protein.

Participants who did not achieve desensitization during the initial or extended phases-defined by a positive OFC-will resume cashew nut protein OIT per the established clinical desensitization protocol implemented at the investigational site, irrespective of their initial randomization group.

Statistical Considerations

An interim analysis is planned once 70% of participants have completed the primary outcome assessment. This analysis will be conducted by an independent Data Monitoring Committee (DMC) to ensure participant safety and evaluate preliminary efficacy signals. Statistical inference during interim analysis will be controlled using appropriate alpha-spending functions to maintain the overall Type I error rate.

ELIGIBILITY:
Inclusion Criteria:

* Cashew nut allergy confirmed prior to the initiation of immunotherapy
* Completion of the first phase of the study, including achievement of the maintenance dose (1200 mg of cashew nut protein) during immunotherapy
* Provision of informed consent for participation in the study
* Adequate cooperation from the patient and/or their legal guardians

Exclusion Criteria:

* Severe asthma
* Poorly controlled mild-to-moderate asthma, defined as:

  * FEV1 < 80% (below the 5th percentile),
  * FEV1/FVC ratio < 75% (below the 5th percentile),
  * Hospitalization due to asthma exacerbation within the past 12 months
* Oral, sublingual, or subcutaneous immunotherapy for other allergens during the first year/season of therapy
* Eosinophilic gastrointestinal disorders
* Severe, recurrent episodes of anaphylaxis within the last 6 months
* Chronic illnesses requiring ongoing treatment, including:

  * Cardiac conditions
  * Epilepsy
  * Metabolic disorders
  * Diabetes mellitus
* Use of the following medications:

  * Daily oral corticosteroid therapy >1 month within the past 12 months
  * At least two courses of oral corticosteroids (minimum duration of 7 days each) in the past 12 months
  * One course of oral corticosteroids (minimum 7 days) within the past 3 months
  * Biologic therapies
  * Treatment with β-blockers, ACE inhibitors, or calcium channel blockers
* Pregnancy
* Lack of informed consent for participation
* Lack of cooperation from the patient

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Sustained unresponsiveness determined by the outcome of the OFC | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Percentage of patients achieving sustained unresponsiveness after 1200 mg cashew nut protein oral immunotherapy, defined as tolerating 4 g of cashew nut powder in OFC after 4 weeks of cashew nut avoidance.

SECONDARY OUTCOMES:
Changes in cashew nut protein tolerance during OFC | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Comparison of the amount of cashew nut protein tolerated during each oral food challenge (OFC) by each patient. Every OFC will be performed according to PRACTALL guidelines.
Adverse event | 11 months on the maintenance dose of OIT (±3 weeks) and a 4 week break (+/- 7 days).
  Quantity and severity of adverse effect divided into 3 categories: mild, moderate and severe reactions.
Quality of life - FAQLQ (Food Allergy Quality of Life Questionnaire) | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Assessment of the quality of life of patients and their families before each open oral cashew nut protein challenge trial (impact of allergy on family life) based on the Food Allergy Quality of Life Questionnaire (FAQLQ). Based on the FAQLQ score, quality of life will be assessed on a scale ranging from minimal to severe impairment due to food allergy.
Basophil activation test (BAT) | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Assessment of CD63+ basophil marker expression prior to desensitisation and before any OFC.
Evaluation of Predictive Factors for the Acquisition of Sustained Unresponsiveness - wheal diameter in PTS | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  The following parameters will be assessed: Wheal diameter in PTS after exposure to cashew nut powder and cashew nut, measured in millimeters (mm). All outcomes will be measured before OIT, before the 4-week break, and after the 4-week break during OIT.
SIgE (specific immunoglobulin E) (kUA/l) levels | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Difference in sIgE (specific immunoglobulin E) (kUA/l) levels against cashew, walnut, pistachio, peanut, hazelnut and almond allergens, all outcomes will be measured before OIT, before the 4-week break, and after the 4-week break during OIT.
Air condensate | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Evaluation of pro-inflammatory cytokine levels in exhaled air condensate
Evaluation of Predictive Factors for the Acquisition of Sustained Unresponsiveness | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  The following parameters will be assessed: sIgE (specific immunoglobulin E) (kUA/l) levels against cashew, sIgG4 (immunoglobulin IgG4) (mgA/l) levels against cashew, and the result of the basophil activation test (BAT) against cashew. All outcomes will be measured before OIT, before the 4-week break, and after the 4-week break during OIT.
IgG4 (immunoglobulin IgG4) (mgA/l) levels | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Difference in sIgG4 (immunoglobulin IgG4) (mgA/l) levels against cashew, walnut, pistachio, peanut, hazelnut and almond allergens, all outcomes will be measured before OIT, before the 4-week break, and after the 4-week break during OIT.
Cut-off Values for Sustained Unresponsiveness Prediction - PTS wheal diameter | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Identification of the PTS wheal diameter measured in millimeters (mm) above which the patient is unlikely to achieve sustained unresponsiveness as a result of immunotherapy.
Cut-off Values for Sustained Unresponsiveness Prediction - sIgE | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Identification of the concentrations of specific IgE to cashew nut (kUA/L) levels, above which the patient is unlikely to achieve sustained unresponsiveness as a result of immunotherapy.
Determination of Threshold Differences Predictive of Sustained Unresponsiveness - PTS wheal diameter | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Identification of the threshold value for the change in PTS wheal diameter measured in millimeters (mm) before and after OIT, that best distinguishes patients who will achieve sustained unresponsiveness from those who will not.
Determination of Threshold Differences Predictive of Sustained Unresponsiveness - sIgE | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Identification of the threshold value for the change in specific IgE to ]cashew nut (kUA/L) levels before and after OIT, that best distinguishes patients who will achieve sustained unresponsiveness from those who will not.
Evaluation of the Impact of Dose Escalation Duration on OIT Efficacy | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Assessment of how the duration of the dose escalation phase during oral immunotherapy (OIT) impacts treatment effectiveness, measured by the number of patients achieving desensitization and/or sustained unresponsiveness.
Predictive Markers of Severe Allergic Reactions - sIgE | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Evaluation of specific IgE levels to cashew nut ( kUA/L) to assess predictive markers of severe allergic reactions.
Predictive Markers of Severe Allergic Reactions - BAT | After 11 months on the maintenance dose of OIT (±3 weeks) and/or a 4-week break (±7 days).
  Evaluation of the basophil activation test (BAT) results (measured by %CD3+) to assess predictive markers of severe allergic reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elizur A, Appel MY, Nachshon L, Levy MB, Epstein-Rigbi N, Koren Y, Holmqvist M, Porsch H, Lidholm J, Goldberg MR. Cashew oral immunotherapy for desensitizing cashew-pistachio allergy (NUT CRACKER study). Allergy. 2022 Jun;77(6):1863-1872. doi: 10.1111/all.15212. Epub 2022 Jan 15. PMID 35000223
- [Background] Wang F, Robotham JM, Teuber SS, Tawde P, Sathe SK, Roux KH. Ana o 1, a cashew (Anacardium occidental) allergen of the vicilin seed storage protein family. J Allergy Clin Immunol. 2002 Jul;110(1):160-6. doi: 10.1067/mai.2002.125208. PMID 12110836
- [Background] Robotham JM, Wang F, Seamon V, Teuber SS, Sathe SK, Sampson HA, Beyer K, Seavy M, Roux KH. Ana o 3, an important cashew nut (Anacardium occidentale L.) allergen of the 2S albumin family. J Allergy Clin Immunol. 2005 Jun;115(6):1284-90. doi: 10.1016/j.jaci.2005.02.028. PMID 15940148
- [Background] Borres MP, Sato S, Ebisawa M. Recent advances in diagnosing and managing nut allergies with focus on hazelnuts, walnuts, and cashew nuts. World Allergy Organ J. 2022 Apr 11;15(4):100641. doi: 10.1016/j.waojou.2022.100641. eCollection 2022 Apr. PMID 35493774
- [Background] Brough HA, Caubet JC, Mazon A, Haddad D, Bergmann MM, Wassenberg J, Panetta V, Gourgey R, Radulovic S, Nieto M, Santos AF, Nieto A, Lack G, Eigenmann PA. Defining challenge-proven coexistent nut and sesame seed allergy: A prospective multicenter European study. J Allergy Clin Immunol. 2020 Apr;145(4):1231-1239. doi: 10.1016/j.jaci.2019.09.036. Epub 2019 Dec 20. PMID 31866098
- [Background] Washio K, Nakamura M, Sato N, Hori M, Matsubara K, Ogura K, Oda Y, Fukunaga A, Yagami A, Matsunaga K. Anaphylaxis in a pectin- and cashew nut-allergic child caused by a citrus bath. Allergol Int. 2022 Jan;71(1):155-157. doi: 10.1016/j.alit.2021.07.006. Epub 2021 Aug 2. No abstract available. PMID 34353728
- [Background] van der Valk JP, Gerth van Wijk R, Dubois AE, de Groot H, Reitsma M, Vlieg-Boerstra B, Savelkoul HF, Wichers HJ, de Jong NW. Multicentre Double-Blind Placebo-Controlled Food Challenge Study in Children Sensitised to Cashew Nut. PLoS One. 2016 Mar 11;11(3):e0151055. doi: 10.1371/journal.pone.0151055. eCollection 2016. PMID 26967158
- [Background] Pajno GB, Fernandez-Rivas M, Arasi S, Roberts G, Akdis CA, Alvaro-Lozano M, Beyer K, Bindslev-Jensen C, Burks W, Ebisawa M, Eigenmann P, Knol E, Nadeau KC, Poulsen LK, van Ree R, Santos AF, du Toit G, Dhami S, Nurmatov U, Boloh Y, Makela M, O'Mahony L, Papadopoulos N, Sackesen C, Agache I, Angier E, Halken S, Jutel M, Lau S, Pfaar O, Ryan D, Sturm G, Varga EM, van Wijk RG, Sheikh A, Muraro A; EAACI Allergen Immunotherapy Guidelines Group. EAACI Guidelines on allergen immunotherapy: IgE-mediated food allergy. Allergy. 2018 Apr;73(4):799-815. doi: 10.1111/all.13319. Epub 2017 Dec 5. PMID 29205393